CLINICAL TRIAL: NCT05145777
Title: Patients Returning to Work After Acute Coronary Syndrome
Acronym: ACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8334
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; ACS; Return to work; Occupational health; Cardiology; Intensive-care unit
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The literature is quite rich concerning the factors which influence the return to work after acute coronary syndrome. They can be divided into three categories: factors linked to the patient, those linked to the workstation and factors linked to an external intervention. A study published in 1992 evaluated a set of predictive factors for recovery one year after acute coronary syndrome and showed that the proportion of clinical factors accounted for 20%, functional factors for 27% but above all socio-economic factors for 45. %.

On the other hand, there are only a few studies that are interested in the return to work after acute coronary syndrome according to the management in occupational medicine, and in particular the realization or not of a pre-return visit.

The results of a survey published in 2016 show that the recommendations made during the return visit were significantly different depending on whether or not there was a pre-return visit and concerned all types of pathology.

In view of all of these elements, it seems important to the investigators to study the expected benefit of an early orientation towards occupational medicine via the pre-return visit, and to study the factors delaying or favoring the return to work. .

ELIGIBILITY:
Inclusion criteria:

* Age ≥18 years old
* In professional activity during acute coronary syndrome (employee, civil servant, self-employed or looking for a job)
* -Mastering the French language (knowing how to read and write French)
* Agreeing to participate in the study and not having expressed his opposition to the reuse of his data for the purposes of this research

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Inability to provide informed information about the subject (subject in an emergency situation, difficulty in understanding the subject, etc.)
* Subject under safeguard of justice
* Subject under guardianship or guardianship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subject in professional activity during acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Study of the contribution of the pre-return visit to the return to work after acute coronary syndrome | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Marc André GOLTZENE, MD, Principal Investigator — Service de Pathologie Professionnelle - Médecine de Travail - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Pathologie Professionnelle - Médecine de Travail - Hôpitaux Universitaires de Strasbourg, Strasbourg, France